CLINICAL TRIAL: NCT06228924
Title: First-in-Human, Open-Label, Safety, Tolerability, Dose-Finding, Pharmacodynamic and Cardiac Transgene Expression Study of TN-401, a Recombinant Adeno-associated Virus Serotype 9 (AAV9) Containing Plakophilin-2 (PKP2) Transgene, in Adults With PKP2 Mutation-Associated Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC)
Brief Title: Open-label, Dose Escalation Study of Safety and Preliminary Efficacy of TN-401 in Adults With PKP2 Mutation-associated ARVC
Acronym: RIDGE-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tenaya Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TN-401-0012
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: PKP2 Mutation Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC); Arrhythmogenic Cardiomyopathy (ACM); PKP2-associated ARVC; PKP2-ARVC; PKP2-ACM; Adeno Associated Virus (AAV); Gene Therapy; Gene Transfer; Genetic cardiomyopathy; Heart Failure
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Dose for Cohort 1 will be 3E13 vg/kg
  Interventions: Genetic: TN-401
- Cohort 2 (Experimental): Dose for Cohort 2 will be 6E13 vg/kg
  Interventions: Genetic: TN-401

INTERVENTIONS:
Genetic: TN-401 — TN-401 is a recombinant adeno-associated virus serotype 9 (AAV9) gene therapy containing Plakophilin-2 (PKP2) transgene. It is a single (one-time) intravenous dose.

SUMMARY:
This first-in-human study is designed to evaluate the safety, and preliminary efficacy (PD) of TN-401 gene therapy in adult patients with symptomatic PKP2 mutation-associated ARVC.

DETAILED DESCRIPTION:
The RIDGE-1™ open-label Safety, Tolerability, Dose-finding, PD and Cardiac Transgene Expression Study will enroll up to 15 patients in two planned dose cohorts. Patients in each cohort will receive a single intravenous (IV) dose of TN-401. Following Data Safety Monitoring Board (DSMB) review of each dose cohort, the next dose cohort will be initiated. DSMB review will also be needed to expand the dose cohorts. The dose for Cohorts 1/1a will be 3E13 (3 × 1013) vg/kg and the dose for Cohorts 2/2a will be 6E13 (6 × 1013) vg/kg.

ELIGIBILITY:
Inclusion Criteria:

* PKP2 mutation (pathogenic or likely pathogenic)
* Arrhythmogenic Right Ventricular Cardiomyopathy as defined by the 2010 revised Task Force Criteria
* Left Ventricular Ejection Fraction ≥50%
* Functioning Implantable Cardiac Defibrillator with remote integration capabilities at least 9 months prior to Screening
* NYHA Functional Class I, II, or III
* Frequent premature ventricular contractions (PVCs)

Exclusion Criteria:

* Ventricular tachycardia (VT) ablation within 6 months of Screening or planned VT ablation within 6 months after Screening
* High AAV9 neutralizing antibody titer
* Prior myocardial infarction
* Right Ventricular Heart Failure
* Class IV Heart Failure
* Clinically significant renal disease
* Clinically significant liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Number and severity of Adverse Events over the course of the study. | 52 weeks
Number of Serious Adverse Events related to study drug. | 5 years

SECONDARY OUTCOMES:
To assess changes in daily PVC and NSVT counts | Week 52
To assess frequency of ICD therapy administration | Week 52
To assess frequency of sustained VT | Week 52

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.tenayatherapeutics.com/wp-content/uploads/2023-BCVS_PKP2-Novel-Model_Xu.pdf
- See also: Related Info — https://www.tenayatherapeutics.com/wp-content/uploads/PKP2-Gene-Therapy-for-Arrhythmogenic-Right-Ventricular-Cardiomyopathy.pdf
- See also: Related Info — https://www.tenayatherapeutics.com/wp-content/uploads/04152022_PKP2-Presentation_HRS2022_v6.pdf
- See also: Related Info — https://www.tenayatherapeutics.com/wp-content/uploads/Cardiac-AAV9-PKP2-therapy-Abstract-final.pdf